CLINICAL TRIAL: NCT06610318
Title: Brief Strategies for Improving Health Outcomes
Brief Title: Feasibility and Acceptability of a Single Session of Imagery Rescripting in a Community Sample of Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000529
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Feasibility Studies; Acceptability; Depressive Symptoms; Disordered Eating Behaviors
MeSH Terms: conditions — Depression; Disordered Eating Behavior | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Imagery rescripting (Experimental): This condition has three stages. In the first stage, participants were asked to select their most distressing memory related to their appearance (not physical or sexual trauma). They were asked to visualize the selected memory, in detail, as if it were happening to them again. Then, interventionists used a downward arrow technique to identify two-to-three maladaptive core schema. In the second stage, participants were asked to identify a real or imagined trusted adult. Then, they were asked to imagine what their younger self might need to cope with or feel calmer in the situation of their selected memory. In the third stage, the participant was instructed to imagine asking the trusted adult for what they need and to imagine the trusted adult providing their selected interventions and describe how they feel afterwards. These procedures were then repeated with participants' most distressing memory related to eating. This session was remote delivered via Zoom.
  Interventions: Behavioral: imagery rescripting
- Nutrition education control (Active Comparator): The active control condition consisted of a time- and attention-matched general nutrition education session. The curriculum for this intervention included information from the United States Department of Agriculture's Dietary Guidelines (e.g., food labels, describing the benefits of macronutrients). This session was remote delivered using Zoom.
  Interventions: Behavioral: nutrition education

INTERVENTIONS:
Behavioral: imagery rescripting — This condition has three stages. In the first stage, participants were asked to select their most distressing memory related to their appearance (not physical or sexual trauma). They were asked to visualize the selected memory, in detail, as if it were happening to them again. Then, interventionists used a downward arrow technique to identify two-to-three maladaptive core schema. In the second stage, participants were asked to identify a real or imagined trusted adult. Then, they were asked to imagine what their younger self might need to cope with or feel calmer in the situation of their selected memory. In the third stage, the participant was instructed to imagine asking the trusted adult for what they need and to imagine the trusted adult providing their selected interventions and describe how they feel afterwards. These procedures were then repeated with participants' most distressing memory related to eating. This session was remote delivered via Zoom.
  Arms: Imagery rescripting
Behavioral: nutrition education — The active control condition consisted of a time- and attention-matched general nutrition education session. The curriculum for this intervention included information from the United States Department of Agriculture's Dietary Guidelines (e.g., food labels, describing the benefits of macronutrients). This session was remote delivered using Zoom.
  Arms: Nutrition education control

SUMMARY:
Negative experiences related to eating and appearance (NEREAs), such as critical commentary from parents about food, are common. They are also associated with depression and disordered eating, predictors of early mortality. Imagery rescripting (IR) is a therapeutic process during which individuals are guided through recalling distressing memories, like NEREAs, and generating ideas for bringing support into these memories. Single sessions of IR demonstrate promise in shifting the primary negative consequences of NEREAs in clinical samples of women. The current study examined the feasibility and acceptability of a remote-delivered, single session of IR in a community sample of men and women with NEREAs.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. endorse a history of at least one negative experience related to eating and/or appearance

Exclusion Criteria:

1. endorsed a current major medical condition;
2. met criteria for a full threshold psychiatric disorder (of moderate intensity when severity ratings are necessary, such as for substance use disorders and binge eating disorder);
3. were at high risk for suicide;
4. endorsed current or recent pregnancy or anticipated becoming pregnant within the next year;
5. were taking medication known to affect eating, weight and/or chronic disease risk;
6. were participating in eating, weight, or diabetes programming;
7. experienced weight loss > 10% in the past six months; and/or
8. could not complete study procedures in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
enrollment | once, at baseline, over the duration of recruitment to obtain the sample size of interest
  the total number of participants enrolled in the study and a demographic description of these participants, including their sex, gender, race, ethnicity, age and body mass index
fidelity | during the intervention session only
  the % of intervention curriculum the interventionists cover during their intervention session as rated by research staff using a curriculum checklist
data collection completeness | baseline, intervention, 1-month, and 3-month
  % of missing data collected at all study visits
intervention acceptability | these data will be collected during the 1-month follow-up visit
  captured via self-report survey items created by the researchers; participants were asked questions such as the extent to which they liked engaging in the intervention; response options are on a Likert-type scale ranging from strongly agree to strongly disagree; average scores at the item level will be generated by condition
safety | these data will be collected during and between all study visits, from baseline though the 3-month follow-up visit
  frequency of adverse events
retention | from baseline through the 3-month follow-up visit
  the % of participants retained at each visit relative to baseline (i.e., percentage of total enrolled who attended the intervention visit, the 1-month follow-up visit, and the 3-month follow-up visit)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kelly NR, Doty KJ, Schrag BHC, Bryant S, Plezia S, Parr NJ, Budd EL. Feasibility and acceptability of a pilot randomized trial of a single session of imagery rescripting targeting the primary consequences of negative experiences with eating and appearance. Pilot Feasibility Stud. 2025 Apr 23;11(1):51. doi: 10.1186/s40814-025-01630-8. PMID 40270079